CLINICAL TRIAL: NCT06665789
Title: Mindfulness-Based Stress Reduction in Obese Women With Polycystic Ovary Syndrome (PCOS): A Randomized Controlled Trial
Brief Title: Mindfulness-based Stress Reduction in Obese Women With Polycystic Ovary Syndrome (PICOS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Leyla Kaya, Assoc. Prof., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 17.04.2024/34
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Obesity; Polycystic Ovary Syndrome; Stress
Keywords: Emotional Appetite; Polycystic Ovary Syndrome; Obesity; Stress; Cognitive Triad; Mindfulness
MeSH Terms: conditions — Obesity; Polycystic Ovary Syndrome | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single (Participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Mindfulness-based stress reduction training will be given to women selected for the experimental group for 8 weeks.
  Interventions: Behavioral: Mindfulness-based Stress Reduction
- Control (No Intervention): Women in the control group receive routine care at the same hospital's polyclinics.

INTERVENTIONS:
Behavioral: Mindfulness-based Stress Reduction — An 8-week Mindfulness-based stress reduction training programme
  Arms: Experimental

SUMMARY:
The aim of this study was to evaluate the effects of a mindfulness-based stress reduction (MBSR) program on Stress, depression, anxiety, cognitive triad and emotional appetite in obese women with polycystic ovary syndrome (PCOS).

DETAILED DESCRIPTION:
The aim of this study was to evaluate the effects of mindfulness-based stress reduction (MBSR) program on stress, depression, anxiety, cognitive triad and emotional appetite in obese women with polycystic ovary syndrome (PCOS).

This study was designed as a single-blind pilot randomized controlled trial. It is planned to be conducted between November 2024 and January 2025 at Zeynep Kamil Women and Children's Diseases Education and Research Hospital.

Power analysis using G*Power 3.0.10 showed that at least 44 samples were sufficient for 2 groups with Effect size 1. 72, 95% Power and 5% margin of error. Participants to be included in the groups were selected from the sample using a random sampling method with an equal distribution ratio (distribution ratio = 1:1).

Eligible women were randomized into the intervention group (n=22) and the control group (control) (n=22). Women assigned to the intervention group received the MBSR program. MBSR had eight weekly sessions of two hours each and a full-day retreat between the 7th and 8th sessions. The control group received routine care in the hospital but did not receive any other intervention during this period.

The pre-test data of the study were collected by the researcher using a face-to-face interview, a Personal Information Form containing demographic questions, and the measurement tools used in the study. At the end of the 8 weeks, the post-test data were collected using the same method.

The participants were given explanations about the MBSR program and it was stated how, for how long, and where to practice. The online MBSR program was completed by the participants in a way specific to each session (with mind, body, and breathing exercises). The MBSR program was implemented in this way for 8 weeks (eight sessions in total and one session per week). In addition, the participants were given homework (audio recording) to do throughout the week (until the next session) in the form of repeating mindfulness meditation practices. At the end of the eighth week, the measurement tools were re-administered to the participants who attended all eight sessions and completed their homework, and the post-test data were obtained.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18-40
* Body mass index (BMI) ≥ 40 kg/m2
* Women with a diagnosis of polycystic ovary syndrome

Exclusion Criteria:

* Psychiatric illness
* Pregnant women
* Thyroid dysfunction
* Cushing's syndrome
* Hyperprolactinemia
* Cancer history
* Pharmacological treatment for obesity
* Any type of bariatric surgery
* Absence of any psychiatric illness or comorbidities
* Current enrollment in a stress reduction program
* Mindfulness practice within the past 6 months (regular formal practice at least once a week)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Famale
Enrollment: 100 (Actual)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Depression Anxiety Stress Scale (DASS 21) | Imediately after participants are assigned to groups and eight weeks later
  In this scale (DASS-21), there are 7 questions each to measure the dimensions of depression, stress and anxiety. The scale is a 4-point Likert Type Scale; 0 -3. Depression, anxiety and stress scores are measured by summing the scores of the related items. A minimum of 0 and a maximum of 21 points can be obtained in each dimension.
Emotional Appetite Questionnaire (EAQ) | Imediately after participants are assigned to groups and eight weeks later
  In this questionnaire, the presence of emotional eating is assessed in negative/positive emotions (14 items) and situations (8 items). The negative total score is obtained by adding and averaging the scores of negative emotions and negative situations (EAQ), and the positive total score is obtained by adding and averaging the scores of positive emotions and positive situations (EAQ). This scale, which does not have a cut-off score for emotional eating, analyzes the emotions and situations in which emotional eating behavior can occur specifically.
Ruminative Thought Style Questionnaire (RTSQ) | Imediately after participants are assigned to groups and eight weeks later
  It is a 20-item 7-point Likert-type scale (1=does not describe me at all, 7=describes me very well). There is no cut-off score for the scale result. The minimum score can be 20 and the maximum can be 140, and the results only show the tendency for ruminative thinking. As the score increases, it can be said that the person's ruminative thinking style is intense. This scale tries to evaluate the general way of thinking of the person without taking into account the person's current emotional state and without dividing it into subscales. This shows that the scale can be used in all psychopathological disorders. Since it is not related to any psychopathology, the total score does not indicate psychiatric disorders.
Cognitive Triad Inventory | Imediately after participants are assigned to groups and eight weeks later
  In the seven-point Likert-type form consisting of 36 items, one option is marked for each item between "I do not agree at all" (1) and "I completely agree" (7). When scoring the items, all negative items are reverse coded and low scores from the scale reflect the negative cognitive triad, while high scores reflect the positive cognitive triad.

CONTACTS AND LOCATIONS:
Overall Officials: Leyla Kaya, PhD, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Zeynep Kamil Women and Children's Diseases Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No